CLINICAL TRIAL: NCT05283070
Title: Comparing Patient Reported Outcomes to Objective Measures of Function in Patients With Chronic Pain: Using the 2 Minute Walk Test and Elevation and Movement Lift Test, and Heart Rate Variability
Brief Title: Correlating Heart Rate Variability and Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Canadian Forces Health Services Centre Ottawa (Other)
Responsible Party: Principal Investigator, Gaurav Gupta, Principal Investigator, Canadian Forces Health Services Centre Ottawa
Other Study IDs: 2020-044
Record Dates: First submitted 2022-02-12; First posted 2022-03-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Volunteers without preexisting chronic pain and/or mental health issues
  Interventions: Other: Questionnaires, physical tests, and heart rate variability measures
- Patients with chronic pain: Patients with chronic pain and/or mental health issues
  Interventions: Other: Questionnaires, physical tests, and heart rate variability measures

INTERVENTIONS:
Other: Questionnaires, physical tests, and heart rate variability measures — The 2MWT will be conducted in an unobstructed hallway with patients being asked to walk at moderate intensity (brisk walk) for the duration of the activity (2 minutes). The amount of distance in metres will be recorded.
  The EMLi movement consists of pushing a 2kg weighted ball from the chest level forward, and then raising the ball overhead, before returning it to the starting position (Figure 1). The number of repetitions done at moderate intensity will be recorded after 60 seconds.
  HRV and questionnaires previously listed

SUMMARY:
The Canadian Armed Forces (CAF) has limited data on baseline quality of life measures and objective measures of function, for active serving members with chronic pain. This study aims to collect this data using patient reported outcomes and 2 minute walk test (2MWT) while validating the newly created Elevation Movement Lift Off Test (EMLi) and correlating the data with heart rate variability (HRV) while comparing performance to healthy controls

DETAILED DESCRIPTION:
Objective The Canadian Armed Forces (CAF) has limited data on baseline quality of life measures and objective measures of function, for active serving members with chronic pain. This study aims to collect this data using patient reported outcomes and 2 minute walk test (2MWT) while validating the newly created Elevation Movement Lift Off Test (EMLi) and correlating the data with heart rate variability (HRV) while comparing performance to healthy controls.

Procedure Patients will complete pre-defined questionnaires on their pain condition, potential risk factors, and function. This data includes information on demographics, occupation, pain conditions and its impact on life, exercise levels, mood, childhood experiences, views on your condition and requests for care support. For patients and controls investigators will collect performance and heart rate measures while at rest, walking and lifting tests.

Risks and Mitigation Strategies Participation in this study is voluntary and volunteers can withdraw consent at any time without having any effect on access to future medical care.

Due to the nature of this study there are no significant associated risks. Any patients developing issues consistent with cardiopulmonary compromise will be treated according to the standard of care, stabilized and referred on for further evaluation.

The data collected will be stored in a locked Protected-B cabinet at the Canadian Forces Health Services Centre only and access will be restricted to the research team. The spreadsheet generated from this data will be password protected and anonymized. Only the research team will have access to this data.

The data intake protocol included completing a questionnaire with:

1. Demographics - age, gender, rank, working status, medical category
2. Height and weight, waist to hip ratio
3. Medications in the following groups

   1. Antipsychotics
   2. Antihypertensives
   3. Antidepressants
   4. Oral Contraceptive Pill
   5. Stimulants
   6. Cannabinoids
4. Activity and Food Intake

   a. Alcohol, caffeine, energy drinks, food, intense exercise, tobacco, cannabis
5. Patient Reported Outcomes at baseline (Appendix B)

   1. Body Pain Diagram
   2. Pain, Enjoyment and General Activity Scale (PEG)
   3. Pain Disability Index
   4. Hospital Anxiety and Depressions Scale (HADS)
   5. Adapted Deployment Risk & Resilience Inventory 2 Section J: Unit Support Exercise Questionnaire
   6. Brief Trauma Questionnaire (BTS)
   7. Litigation Status

The physical activity measures to be taken are:

1. 2 minute walk test (2MWT)
2. Elevation & Movement Lift test (EMLi)
3. Heart rate variability and Vagal Tone (VT) indices (12 minutes total) - Firstbeat Bodyguard 2 (Firstbeat Finland)

   1. Supine (3 minutes)
   2. Sit (3 minutes)
   3. Stand (3 minutes)
   4. 2MWT (2 minutes)
   5. EMLI (1 min)
4. Borg Perceived Exertion Scale

Sample Size Calculation Current studies on chronic pain and HRV ranged from samples sizes of 12-731 patients and 11-1633 controls showing a standard mean difference of 0.15 to 73.6 depending on the variable and condition being studied. Quintana described an analysis of 297 HRV effect sizes from between-group/case-control studies and concluded that for HRV studies a sample size of 233, 61, and 21 participants are required, respectively, to detect small, medium and large effect sizes, respectively. The Laborde et al. guidelines for HRV and VT research rely on this estimation and therefore investigators have selected a sample of 100 patients with chronic pain and 50 controls .

Statistical analysis The difference in performance during the upper and lower repetition tests will be evaluated between the groups. This includes vagal tone measures/ heart rate variability, number of repetitions and perceived exertion. This will be evaluated using multiple ANOVA tests, corrected for multiple comparisons using the Games-Howell post-hoc test.

Correlation analysis between selected variables will be done using multiple Pearson correlations, and adjusted for multiple comparisons using the Benjamini-Hochberg false discovery rate equation.

Acquisition of electrocardiogram data (ECG) data will be via a HRV capture device with data sampled at 1000 Hz. Disposable electrodes will be placed on the participant chest (Bodyguard) or ear (EM Wave Pro Plus). Only one device will be used for all patients in the study as each device is currently being vetted by the research team. The electrodes will be positioned in accordance to the device use guidelines. When needed, the skin will be prepared, in order to improve signal quality (cleaning or hair removal). The ECG sampling rate of 1000 Hz, which is consistent with the more conservative guidelines.The participant may be asked to sit quietly for 5 minutes prior to data collection and then deep breath in and out for 1 minute.

VT Analysis HRV data will be visually inspected and edited off-line with CardioEdit software (Brain-Body Center, the University of Illinois at Chicago). HRV and VT indices will be calculated using CardioBatch Plus software (Brain-Body Center for Psychophysiology and Bioengineering, the University of North Carolina at Chapel Hill, 2016) consistent with procedures developed by Prof. Porges. The edited heart period sequences were analyzed with specific algorithms developed to quantify three metrics of respiratory sinus arrhythmia (RSA): Porges-Bohrer time domain method (RSAP-B), peak-to-trough (P2T), and the accumulated variances across a high frequency band (HF) from the spectral analyses.

Vagal efficiency will be calculated by the slope between the dynamic and synchronous shifts in RSA and heart period, which provides a measure of regulation of heart rate by vagal pathways.

ELIGIBILITY:
Inclusion Criteria:

* for patients male and female between 18 and 60 years old
* seen within the CFO-P
* diagnosed with one or more chronic pain condition

Exclusion Criteria:

* adults who are unable to give their own consent
* adults with uncontrolled mental health issues For Controls
* Pacemaker/Cardiac Issues
* SSRI/Beta Blocker/Anticholinergic medication use in controls
* Migraine, cold medication, antihistamine, drugs use (ie cannabis <48hours)

Patients/controls will be asked

* to bring exercise attire including running shoes,
* not to drink alcohol within 24 hours of testing,
* not to consume caffeinated products (ie energy drinks or tea/coffee) within 2 hours of the testing,
* not to eat within 2 hours of testing,
* not to participate in intense exercise for 24 hours before testing,
* not to use nicotine products (smoke, vaping, and tobacco) in the 2 hours before testing,
* not to use plant-based cannabis products 2 hours before testing
* to use the bathroom before testing.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: A convenience sample of 100 patients with chronic pain and 50 pain-free controls will be asked to complete the research protocol (see sample size calculation below). Our study population will be Canadian Forces members between the ages of 18-60 years old, suffering from chronic pain, seen within the CFO-P. Controls will be recruited from Canadian Forces bases in Ottawa, Borden and/or Petawawa.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | baseline
  Both sympathetic and parasympathetic nervous systems are involved in regulating pain states and may be disturbed in chronic pain. This disruption of the autonomic nervous system may be measured by variability of the interval between consecutive heart beats

SECONDARY OUTCOMES:
2 minute walk test (2MWT) | baseline
  how far someone can walk in 2 minutes
Elevation & Movement Lift test (EMLi) | baseline
  how many repetitions in 1 minute
Pain, Enjoyment and General Activity Scale (PEG) | baseline
  Pain, Enjoyment and General Activity Scale (PEG) which is a 3-question scale with scores from 0-10 looking to describe the change (if any) in activity limitations, symptoms, emotions and overall quality of life, related to the pain condition. Higher scores indicate poorer pain and function.
The Pain Disability Index (PDI) | baseline
  a 7-item questionnaire to investigate the magnitude of self-reported pain-related disability, independent from region of pain or pain-related diagnosis. The items of the questionnaire are assessed on a 0-10 numeric rating scale in which 0 means no disability and 10 is maximum disability

CONTACTS AND LOCATIONS:
Locations (1):
- Canadian Forces Health Services Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No